CLINICAL TRIAL: NCT04910620
Title: The Evaluation of TCI378 and TCI507 Probiotics on Weight-lowering Efficacy in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201912029RSA
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Weight Reduction
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo without TCI378 and TCI507
  Interventions: Drug: Placebo
- TCI378 (Experimental): probiotics TCI378 (Lactobacillus plantarum TCI378)
  Interventions: Drug: TCI378
- TCI507 (Experimental): TCI507 (Lactobacillus plantarum TCI507)
  Interventions: Drug: TCI507

INTERVENTIONS:
Drug: Placebo — Placebo only
  Arms: Placebo
Drug: TCI378 — TCI378 (Lactobacillus plantarum TCI378)
  Arms: TCI378
Drug: TCI507 — TCI507 (Lactobacillus plantarum TCI507)
  Arms: TCI507

SUMMARY:
Obesity is a serious global public health issue. Many reports have showed that the use of appropriate probiotics can bring benefits to the health of the host and promote the balance of gut microbiota. Clinical experimental data show that the supplement of probiotics can help regulate gut function and weight control, and etc.

TCI378 (Lactobacillus plantarum TCI378) is a probiotic extracted from Korean kimchi, and TCI507 (Lactobacillus plantarum TCI507) is a probiotic extracted from the oranges peels. These two strains of probiotics have been verified by in vitro experiments to have the effect of hydrolyzing bile salts, inhibition of the production of fat cells. Therefore, we want to evaluate whether the probiotics TCI308 and TCI507 have effects on reduction of body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 20 and 65 who are willing to sign the consent form of the subject.
2. For those with BMI ≥ 24, men's body fat ≥ 25%, women's body fat ≥ 30%
3. Those who are not pregnant and are willing to cooperate with contraception during the trial period.
4. Those who have no history of cardiovascular disease, organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine disease, mental disease, alcohol or drug abuse, and other major organic diseases (according to medical history).

Exclusion Criteria:

1. Pregnant women, people with a history of cardiovascular disease, organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine diseases, mental illness, alcohol or drug abuse, and other major organic diseases (according to medical history).
2. Those who had undergone major surgery or bariatric surgery (according to medical history).
3. Currently or within 3 months before participating in the screening, those subjects used drugs that can affect body fat or increase weight significantly, such as systemic corticosteroids, tricyclic antidepressants, atypical psychiatric drugs, and mood stability Drugs (according to medical history).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2024-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether the probiotics TCI378 (Lactobacillus plantarum TCI378) and TCI507 (Lactobacillus plantarum TCI507) have effect on reduction of body weight. | 8 weeks